CLINICAL TRIAL: NCT02150434
Title: Evaluation of Automatic Oxygen Flow Titration During Walking in Patients With COPD
Acronym: FreeO2rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Canada Foundation for Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FreeO2-Rehab-1
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: COPD; Exercise; Endurance Shuttle Walking Test (Exercise at 85% of Maximal Shuttle Walking Test)
Keywords: Oxygen therapy; Hypoxemia; COPD; Closed-loop; Automated titration,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Hypoxia | interventions — Compressed Air; Air; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Compressed Air (Sham Comparator): compressed air delivered at a fixed flow of 2 L/min
  Interventions: Drug: Compressed air
- Oxygen constant flow (Active Comparator): oxygen delivered at a fixed flow of 2L/min
  Interventions: Drug: Oxygen constant flow
- Automated oxygen titration (Experimental): oxygen at a variable flows delivered by the FreeO2
  Interventions: Device: Automated oxygen titration

INTERVENTIONS:
Device: Automated oxygen titration — Automated oxygen titration every second to maintain stable SpO2 at a predefined value (94% in the present study)
  Other Names: FreeO2 system TM, Oxy'nov.inc
  Arms: Automated oxygen titration
Drug: Compressed air — compressed air delivered at a fixed flow of 2 L/min
  Other Names: Air
  Arms: Compressed Air
Drug: Oxygen constant flow — oxygen delivered at a fixed flow of 2L/min
  Other Names: Oxygen
  Arms: Oxygen constant flow

SUMMARY:
The aim of the current study was to evaluate a new system (FreeO2) that automatically titrates oxygen flow to maintain stable SpO2, in patients with moderate or severe chronic obstructive pulmonary disease during exercise. The investigators hypothesized that continuous automatic adjustment of the oxygen flows during exercise would better maintain patients within the oxygenation target, reduce episodes of desaturation and hyperoxia and would improve walking exercise tolerance in comparison with fixed levels of low-flow oxygen and with compressed air breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years
* Moderate to severe COPD according to the Global Initiative for Chronic Obstructive Lung Disease guidelines
* Who did not require long-term oxygen therapy were included in the study.
* Patients were also selected on the basis of known (end-exercise SpO2 < 90% on a previous exercise test) or suspected (SpO2 < 95% at rest) desaturation during exercise

Exclusion Criteria:

* Episode of exacerbation or hospitalisation within last four weeks
* Current medical condition that could influence exercise tolerance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time within predefined SpO2 target | during exercise (Endurance shuttle walking test)
  The primary outcome of the study was the percentage of exercise time during which patients were kept within the SpO2 target of 92 to 96%

SECONDARY OUTCOMES:
Exercise tolerance | duration of ESWT
  Endurance shuttle walking test time and distance

OTHER OUTCOMES:
Physiological parameters | during ESWT
  Physiological parameters continuously recorded by the FreeO2 system (SpO2, end-tidal CO2 [EtCO2], respiratory rate, heart rate and oxygen flow when automated oxygen titration was activated), blood gases (before and after ESWT and after recovery) and dyspnea assessment during ESWT with a 10-point Borg scale

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, MD PhD, Principal Investigator — Centre de recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Québec
Locations (1):
- Centre de recherche de l'IUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080